CLINICAL TRIAL: NCT02807285
Title: An Open Label, MultiCenter, Expanded-Access Program for Ocrelizumab in Patients With Primary Progressive Multiple Sclerosis
Brief Title: Expanded Access Program for Ocrelizumab in Participants With Primary Progressive Multiple Sclerosis
Status: No longer available | Type: Expanded Access
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29972
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Participants will receive 600 mg ocrelizumab as two 300 mg infusions separated by 14 days, every 24 weeks.
  Other Names: RO4964913

SUMMARY:
The primary objective of this expanded access program is to provide ocrelizumab as treatment for eligible participants with primary progressive multiple sclerosis (PPMS) before it is commercially available in the United States (U.S.) for the indication of PPMS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years (inclusive)
* Diagnosis of PPMS in accordance with the revised 2010 McDonald criteria and the presence or documented history of cerebrospinal fluid oligoclonal bands by isoelectric focusing or elevated immunoglobulin G (IgG) index
* Expanded Disability Status Score (EDSS) of 2.0 to 6.5 points at screening
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of less than (<)1 percent (%) per year during the treatment period and for at least 24 weeks after the last dose of study treatment or until their B-cells have repleted, whichever is longer

Exclusion Criteria:

* History of relapsing-remitting multiple sclerosis (RRMS), progressive relapsing multiple sclerosis (PRMS) or secondary progressive multiple sclerosis (SPMS) at screening
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History or known presence of recurrent or chronic infection
* History of recurrent aspiration pneumonia requiring antibiotic therapy
* History of cancer, including solid tumors and hematological malignancies (except basal cell, in situ squamous cell carcinomas of the skin, and in situ carcinoma of the cervix of the uterus that have been excised and resolved with documented clean margins on pathology)
* History of or currently active primary or secondary immunodeficiency
* History of coagulation disorders because ocrelizumab is administered via infusion
* Known presence or history of other neurologic disorders
* Significant, uncontrolled disease, such as cardiovascular (including cardiac arrhythmia), pulmonary (including chronic obstructive pulmonary disease), renal, hepatic, endocrine, gastrointestinal, or any other significant disease
* Congestive heart failure
* Known active bacterial, viral, fungal, mycobacterial infection, or other infection
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the expanded access program (EAP)
* Contraindications for or intolerance to oral or IV corticosteroids, including IV methylprednisolone
* Treatment with therapies approved for relapsing forms of Multiple Sclerosis (MS), including: Beta interferons, glatiramer acetate, fingolimod (Gilenya®), teriflunomide (Aubagio®), dimethyl fumarate (Tecfidera®), IV immunoglobulin, plasmapheresis, or other immunomodulatory therapies within 12 weeks prior to enrollment (Participants should not be excluded from the EAP due to previous treatment with rituximab)
* Participants who have received fingolimod (Gilenya®) or dimethyl fumarate (Tecfidera®) if their lymphocyte count is not within normal values
* Previous treatment with natalizumab (Tysabri®) within 6 months of screening (Participants are not eligible for the EAP if they have been treated with natalizumab (Tysabri) for more than 1 year)
* Any previous treatment with alemtuzumab (Lemtrada®)
* Any previous or current treatment with any experimental procedure for MS

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (56):
- United States (56):
  - Phoenix Neurological Associates Ltd, Phoenix, Arizona
  - Territory Neurology and Research Institute, Tucson, Arizona
  - Mercy Medical Group; MS Centre Nurse, Carmichael, California
  - Scripps Clinic, La Jolla, California
  - MS Center of Southern California, Newport Beach, California
  - Stanford University, Palo Alto, California
  - Neuro-Therapeutics Inc., Pasadena, California
  - UCSF- Multiple Sclerosis Centre; Department of Neurology, San Francisco, California
  - University Of Colorado, Aurora, Colorado
  - Advanced Neurology of Colorado, LLC, Fort Collins, Colorado
  - Associated Neurologists of Southern CT PC, Fairfield, Connecticut
  - Neurology Associates, Norwich, Connecticut
  - University of Miami Miller School of Medicine; Clinical Reseach Building, Miami, Florida
  - Neurological Services of Orlando, Orlando, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - University of South Florida, Tampa, Florida
  - MS Center of Vero Beach, Vero Beach, Florida
  - Consultants in Neurology Ltd, Northbrook, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Neurology Services, Louisville, Kentucky
  - Steward St. Elizabeth's Medical Center, Boston, Massachusetts
  - Wayne State Uni /Detroit Medical Center, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - The Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - South Shore Neurologic Associates P.C., Patchogue, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center; Department of Neurology, Columbus, Ohio
  - Neurology and Neuroscience Assoc., Inc., Westerville, Ohio
  - Oklahoma Medical Research Foundation; MS Center of Excellence, Oklahoma City, Oklahoma
  - Providence Multiple Sclerosis Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - The Neurology Foundation, Inc., Providence, Rhode Island
  - Sibyl Wray MD Neurology PC, Knoxville, Tennessee
  - Advanced Neurosciences Institute, Nashville, Tennessee
  - University Of Texas Health Science Center Houston, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Neurology Center of San Antonio, San Antonio, Texas
  - University of Vermont, Burlington, Vermont
  - Neurological Associates Inc; Clinical Research, Richmond, Virginia
  - Swedish Neuroscience Institute; Multiple Sclerosis Center, Seattle, Washington
  - Multicare Neuroscience Center of Washington, Tacoma, Washington
  - Columbia St. Mary's Hospital System, Milwaukee, Wisconsin